CLINICAL TRIAL: NCT02150642
Title: Probing Neural Circuitry for the Control of Movement
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-11/2004 / PB_2016-00229
Record Dates: First submitted 2014-05-14; First posted 2014-05-30 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Neurological Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neurological Injury
- No Neurological Injury

SUMMARY:
The investigators are interested in examining 1) the basic organization of spinal and cortical circuitry for the control of movement and 2) the influence of injury of these circuits. To investigate the neuronal circuitry, the investigators use various types of mechanical or electrical stimulation of the limbs, transcranial magnetic stimulation of the cortex and galvanic vestibular stimulation in both uninjured human subjects and subjects with a neurological injury (such as spinal cord injury, or Parkinsons's disease).

ELIGIBILITY:
Inclusion Criteria:

* control subjects: no neurological movement disorder
* patients: neurological movement disorder

Exclusion Criteria:

patients and control subjects:

* presence of any central psychiatric disorder that precludes subject from giving informed and voluntary consent
* presence of any cardiovascular conditions or limitations that restrict the ability to walk on a treadmill continuously for more than 20 minutes
* for the electrical stimulation examination, subjects with metal implants are also excluded
* for the TMS and GVS examination, subjects with the following conditions are excluded: metal implants in the head, cardiac pacemakers, history of migraine headaches, history of major head injury, history of stroke, history of seizures, previous brain neurosurgery, unstable medical conditions, major psychiatric disorders, pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: control subjects without neurological movement disorder AND patients with neurological movement disorder
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2004-05; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Spinal reflex activity | one day
  Spinal reflex activity will be assessed by electrical nerve stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland